CLINICAL TRIAL: NCT01488097
Title: An Open Label Multicenter Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of SBC-102 in Adult Subjects With Liver Dysfunction Due to Lysosomal Acid Lipase Deficiency Who Previously Received Treatment in Study LAL-CL01
Brief Title: Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of SBC-102 (Sebelipase Alfa) in Adult Subjects With Lysosomal Acid Lipase Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-CL04
Record Dates: First submitted 2011-11-26; First posted 2011-12-08 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-06

CONDITIONS: Cholesterol Ester Storage Disease (CESD); Lysosomal Acid Lipase Deficiency; LAL-Deficiency
Keywords: Enzyme replacement therapy (ERT); Lysosomal storage disease; Late onset lysosomal acid lipase (LAL) deficiency; Acid cholesteryl ester hydrolase deficiency, type 2; Acid lipase disease; Cholesterol ester hydrolase deficiency; LAL deficiency; LIPA enzyme deficiency
MeSH Terms: conditions — Cholesterol Ester Storage Disease; Wolman Disease; Lysosomal Storage Diseases | interventions — Sebelipase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Sebelipase Alfa (Experimental): Participants were administered sebelipase alfa once weekly (qw) as an intravenous (IV) infusion at the same dose received in Study LAL-CL01 (0.35, 1, or 3 milligrams per kilogram [mg/kg]) for 4 weeks. After the initial 4 qw doses, participants transitioned to dosing every other week (qow) at either 1 mg/kg (participants who initiated treatment at 0.35 or 1 mg/kg qw) or 3 mg/kg (participants who initiated dosing at 3 mg/kg qw). Subsequent modifications to the dose and dosing frequency were permitted for individual participants based on observed safety, tolerability, and clinical response to treatment. Participants could continue to receive treatment with sebelipase alfa for up to 5 years.
  Interventions: Drug: sebelipase alfa

INTERVENTIONS:
Drug: sebelipase alfa — Sebelipase alfa is a recombinant human lysosomal acid lipase.
  Other Names: SBC-102; Kanuma®

SUMMARY:
This was an extension study to Study LAL-CL01 (NCT01307098). The primary objective of the study was to evaluate the long-term safety and tolerability of sebelipase alfa in participants with liver dysfunction due to lysosomal acid lipase (LAL) deficiency.

DETAILED DESCRIPTION:
Participants who successfully received all 4 doses of sebelipase alfa in Study LAL-CL01 and opted to continue treatment in the extension study underwent screening assessments to determine study eligibility. Eligible participants initiated treatment in the extension study at least 4 weeks after their last dose of sebelipase alfa in Study LAL-CL01. This extension study consisted of a treatment period of up to 5 years, and a follow-up period of approximately 30 days after the last dose of sebelipase alfa.

Cholesteryl ester storage disease (CESD) is the late onset phenotype for LAL deficiency, a lysosomal storage disorder, which also has an early onset phenotype that primarily affects infants. CESD can present in childhood but often goes unrecognized until adulthood when the underlying pathology is advanced. Many of the signs and symptoms are common to patients with other liver conditions.

CESD is an autosomal recessive genetic condition and is characterized by hepatomegaly, persistently abnormal liver function tests (LFTs) and type II hyperlipidemia. Splenomegaly and evidence of mild hypersplenism may affect some patients. Untreated, CESD may lead to fibrosis, cirrhosis, liver failure and death.

ELIGIBILITY:
Inclusion Criteria:

* Participant received all 4 scheduled doses of sebelipase alfa in Study LAL-CL01 with no life-threatening or unmanageable study drug toxicity.

Exclusion Criteria:

* Clinically significant concurrent disease, serious inter-current illness, concomitant medications or other extenuating circumstances
* Clinically significant abnormal values on laboratory screening tests, other than LFTs or lipid panel tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (5):
  - Eureka, California
  - Sacramento, California
  - San Francisco, California
  - Minneapolis, Minnesota
  - New York, New York
- Greater Sudbury, Ontario, Canada
- Prague, Czechia
- Paris, France
- United Kingdom (2):
  - Leeds
  - Salford

REFERENCES:
- [Result] Balwani M, Breen C, Enns GM, Deegan PB, Honzik T, Jones S, Kane JP, Malinova V, Sharma R, Stock EO, Valayannopoulos V, Wraith JE, Burg J, Eckert S, Schneider E, Quinn AG. Clinical effect and safety profile of recombinant human lysosomal acid lipase in patients with cholesteryl ester storage disease. Hepatology. 2013 Sep;58(3):950-7. doi: 10.1002/hep.26289. Epub 2013 Mar 28. PMID 23348766
- [Derived] Malinova V, Balwani M, Sharma R, Arnoux JB, Kane J, Whitley CB, Marulkar S, Abel F. Sebelipase alfa for lysosomal acid lipase deficiency: 5-year treatment experience from a phase 2 open-label extension study. Liver Int. 2020 Sep;40(9):2203-2214. doi: 10.1111/liv.14603. Epub 2020 Aug 9. PMID 32657505
- See also: Alexion website — http://alexion.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants who completed Study LAL-CL01 (received all 4 doses of sebelipase alfa) were screened for eligibility for enrollment in this extension study (LAL-CL04). 8 participants met all enrollment criteria and were enrolled. 1 participant who required a liver transplant no longer met the entry criteria.
Period: Overall Study
Arm/Group | Open-Label Sebelipase Alfa
Started | 8
Received Study Drug in Extension Study | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All participants who received any amount of study drug in the extension study.
Groups:
- Open-Label Sebelipase Alfa: Participants were administered sebelipase alfa qw as an IV infusion at the same dose received in Study LAL-CL01 (0.35, 1, or 3 mg/kg) for 4 weeks. After the initial 4 qw doses, participants transitioned to dosing qow at either 1 mg/kg (participants who initiated treatment at 0.35 or 1 mg/kg qw) or 3 mg/kg (participants who initiated dosing at 3 mg/kg qw). Subsequent modifications to the dose and dosing frequency were permitted for individual participants based on observed safety, tolerability, and clinical response to treatment. Participants could continue to receive treatment with sebelipase alfa for up to 5 years.
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1
  Czechia | 1
  United States | 3
  United Kingdom | 2
  France | 1

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Reporting TEAEs And IARs
Description: Safety and tolerability of sebelipase alfa was primarily assessed by monitoring the number of participants reporting treatment-emergent adverse events (TEAEs), including serious adverse events, and infusion-associated reactions (IARs). The number of participants who discontinued from the study due to a TEAE is also presented. An IAR was defined as any adverse event that occurred during the 2-hour infusion or within 4 hours after the end of the infusion and was assessed by the investigator as at least possibly related to study drug. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module. TEAEs that occurred after the first dose administration at Week 1 through the End of Study (EOS) are presented. End of study was 30 days (+ 7 days) after the last dose of study drug (at Week 260).
Time Frame: From after first dose administration post-Baseline through EOS during study LAL-CL04
Population: Safety Analysis Set: All participants who received any amount of study drug in the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
Participants
  TEAEs | 8
  Serious TEAEs | 1
  IARs | 2
  TEAEs Leading to Study Discontinuation | 0

2. Secondary Outcome: Changes From Baseline In ALT And AST
Description: Changes from Baseline to Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS for alanine aminotransferase (ALT) and aspartate aminotransferase (AST). Baseline values were defined as the last measurement prior to the first infusion of sebelipase alfa in Study LAL-CL04.
Time Frame: Baseline, Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS
Population: Participants in the Full Analysis Set (FAS) for whom ALT and AST data were available at both Baseline and the indicated post-treatment time point. The FAS included all participants who received at least 1 complete infusion of sebelipase alfa in this study and who had at least 1 post-treatment measurement in this study.
Measure: Mean (Standard Deviation); unit: units (U)/liter (L)
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
units (U)/liter (L)
  ALT Week 12 | -35.9 (19.99)
  ALT Week 24 | -38.1 (24.00)
  ALT Week 52: number analyzed (Participants) | 7
  ALT Week 52 | -40.6 (20.50)
  ALT Week 104 | -42.5 (19.65)
  ALT Week 156 | -29.5 (20.38)
  ALT Week 208: number analyzed (Participants) | 7
  ALT Week 208 | -26.7 (30.58)
  ALT Week 260: number analyzed (Participants) | 5
  ALT Week 260 | -31.6 (21.78)
  ALT EOS: number analyzed (Participants) | 7
  ALT EOS | -26.6 (31.10)
  AST Week 12 | -13.9 (7.02)
  AST Week 24 | -12.4 (11.71)
  AST Week 52: number analyzed (Participants) | 7
  AST Week 52 | -18.6 (12.82)
  AST Week 104 | -11.8 (15.59)
  AST Week 156 | -12.8 (9.95)
  AST Week 208: number analyzed (Participants) | 7
  AST Week 208 | -10.4 (14.86)
  AST Week 260: number analyzed (Participants) | 5
  AST Week 260 | -10.8 (13.70)
  AST EOS: number analyzed (Participants) | 7
  AST EOS | -15.3 (14.27)

3. Secondary Outcome: Changes From Baseline In Liver Volume
Description: Changes in liver volume from Baseline to Week 10 or 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS was assessed by magnetic resonance imaging (MRI). Baseline values were defined as the last measurement prior to the first infusion of sebelipase alfa in Study LAL-CL04. Liver volume was expressed as multiples of normal (MN), where normal is defined as 2.5% of body weight.
Time Frame: Baseline, Week 10 or 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS
Population: Participants in the FAS for whom liver volume data were available at both Baseline and the indicated post-treatment time point. The FAS included all participants who received at least 1 complete infusion of sebelipase alfa in this study and who had at least 1 post-treatment measurement in this study.
Measure: Mean (Standard Deviation); unit: Multiples of Normal (MN)
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
Multiples of Normal (MN)
  Week 10 or 12 | -0.096 (0.0892)
  Week 24 | -0.099 (0.1513)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -0.096 (0.0641)
  Week 104: number analyzed (Participants) | 7
  Week 104 | -0.176 (0.0801)
  Week 156: number analyzed (Participants) | 5
  Week 156 | -0.082 (0.0732)
  Week 208: number analyzed (Participants) | 5
  Week 208 | -0.182 (0.0556)
  Week 260: number analyzed (Participants) | 2
  Week 260 | -0.218 (0.0388)
  EOS: number analyzed (Participants) | 2
  EOS | -0.205 (0.0358)

4. Secondary Outcome: Changes From Baseline In Liver Fat Content
Description: Changes in liver fat content from Baseline to Week 10 or 12, Week 24, Week 52, Week 104, Week 156, Week 208, and Week 260, as assessed by multi-echo gradient-echo MRI. Baseline values were defined as the last measurement prior to the first infusion of sebelipase alfa in Study LAL-CL04.
Time Frame: Baseline, Week 10 or 12, Week 24, Week 52, Week 104, Week 156, Week 208, and Week 260
Population: Participants in the FAS for whom liver fat content data were available at both Baseline and the indicated post-treatment time point. The FAS included all participants who received at least 1 complete infusion of sebelipase alfa in this study and who had at least 1 post-treatment measurement in this study.
Measure: Mean (Standard Deviation); unit: percentage fat fraction
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
percentage fat fraction
  Week 10 or 12: number analyzed (Participants) | 5
  Week 10 or 12 | -2.816 (1.8025)
  Week 24: number analyzed (Participants) | 5
  Week 24 | -2.772 (3.0024)
  Week 52: number analyzed (Participants) | 4
  Week 52 | -3.633 (2.5736)
  Week 104: number analyzed (Participants) | 4
  Week 104 | -4.348 (2.4486)
  Week 156: number analyzed (Participants) | 4
  Week 156 | -3.953 (4.1182)
  Week 208: number analyzed (Participants) | 3
  Week 208 | -4.007 (3.4260)
  Week 260: number analyzed (Participants) | 2
  Week 260 | -0.060 (3.4507)

5. Secondary Outcome: Changes From Baseline In GGT And ALP
Description: Changes from Baseline to Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS for gamma glutamyltransferase (GGT) and alkaline phosphatase (ALP). Baseline values were defined as the last measurement prior to the first infusion of sebelipase alfa in Study LAL-CL04.
Time Frame: Baseline, Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS
Population: Participants in the FAS for whom GGT and ALP data were available at both Baseline and the indicated post-treatment time point. The FAS included all participants who received at least 1 complete infusion of sebelipase alfa in this study and who had at least 1 post-treatment measurement in this study.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
U/L
  GGT Week 12 | -13.6 (28.79)
  GGT Week 24 | -13.8 (24.63)
  GGT Week 52: number analyzed (Participants) | 7
  GGT Week 52 | -14.0 (18.89)
  GGT Week 104 | -22.4 (34.01)
  GGT Week 156 | 0.1 (11.32)
  GGT Week 208: number analyzed (Participants) | 7
  GGT Week 208 | 2.3 (10.13)
  GGT Week 260: number analyzed (Participants) | 5
  GGT Week 260 | -6.0 (12.33)
  GGT EOS: number analyzed (Participants) | 7
  GGT EOS | -4.0 (7.70)
  ALP Week 12 | -15.3 (12.09)
  ALP Week 24 | -18.3 (20.74)
  ALP Week 52: number analyzed (Participants) | 7
  ALP Week 52 | -12.4 (18.78)
  ALP Week 104 | -18.0 (9.68)
  ALP Week 156 | -6.4 (11.81)
  ALP Week 208: number analyzed (Participants) | 7
  ALP Week 208 | -5.9 (16.60)
  ALP Week 260: number analyzed (Participants) | 5
  ALP Week 260 | -14.2 (21.32)
  ALP EOS: number analyzed (Participants) | 7
  ALP EOS | -7.9 (20.82)

6. Secondary Outcome: Changes From Baseline In Serum Lipids
Description: Lipid changes from Baseline to Week 10 or 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS were measured in serum for total cholesterol (Total-C), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), and triglycerides (TG). Baseline values were defined as the last measurement prior to the first infusion of sebelipase alfa in Study LAL-CL04.
Time Frame: Baseline, Week 10 or 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS
Population: Participants in the FAS for whom lipid data were available at both Baseline and the indicated post-treatment time point. The FAS included all participants who received at least 1 complete infusion of sebelipase alfa in this study and who had at least 1 post-treatment measurement in this study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
mg/dL
  Total-C Week 12 | -34.5 (40.50)
  Total-C Week 24 | -59.3 (38.83)
  Total-C Week 52: number analyzed (Participants) | 7
  Total-C Week 52 | -73.9 (54.43)
  Total-C Week 104 | -60.8 (50.82)
  Total-C Week 156 | -36.4 (43.90)
  Total-C Week 208: number analyzed (Participants) | 7
  Total-C Week 208 | 1.1 (93.21)
  Total-C Week 260: number analyzed (Participants) | 5
  Total-C Week 260 | -45.5 (50.85)
  Total-C EOS: number analyzed (Participants) | 7
  Total-C EOS | -21.9 (59.89)
  HDL-C Week 12 | 4.9 (3.95)
  HDL-C Week 24 | 5.7 (6.19)
  HDL-C Week 52: number analyzed (Participants) | 7
  HDL-C Week 52 | 9.0 (7.25)
  HDL-C Week 104 | 6.5 (9.04)
  HDL-C Week 156 | 5.2 (9.50)
  HDL-C Week 208: number analyzed (Participants) | 7
  HDL-C Week 208 | 4.9 (4.91)
  HDL-C Week 260: number analyzed (Participants) | 5
  HDL-C Week 260 | 3.4 (8.96)
  HDL-C EOS: number analyzed (Participants) | 7
  HDL-C EOS | 6.7 (9.02)
  LDL-C Week 12 | -34.1 (37.54)
  LDL-C Week 24 | -68.5 (40.22)
  LDL-C Week 52: number analyzed (Participants) | 7
  LDL-C Week 52 | -78.5 (50.91)
  LDL-C Week 104 | -68.7 (43.11)
  LDL-C Week 156 | -40.8 (38.91)
  LDL-C Week 208: number analyzed (Participants) | 7
  LDL-C Week 208 | -20.5 (66.41)
  LDL-C Week 260: number analyzed (Participants) | 5
  LDL-C Week 260 | -43.4 (44.05)
  LDL-C EOS: number analyzed (Participants) | 7
  LDL-C EOS | -35.0 (42.27)
  TG Week 12 | -18.5 (71.93)
  TG Week 24 | -17.5 (37.62)
  TG Week 52: number analyzed (Participants) | 7
  TG Week 52 | -45.2 (66.91)
  TG Week 104 | -24.0 (84.25)
  TG Week 156 | -11.2 (60.45)
  TG Week 208: number analyzed (Participants) | 7
  TG Week 208 | 5.6 (94.18)
  TG Week 260: number analyzed (Participants) | 5
  TG Week 260 | -4.8 (66.03)
  TG EOS: number analyzed (Participants) | 7
  TG EOS | 15.7 (106.54)

7. Secondary Outcome: Changes From Baseline In Serum Ferritin
Description: Changes from Baseline to Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS for serum ferritin. Baseline values were defined as the last measurement prior to the first infusion of sebelipase alfa in Study LAL-CL04.
Time Frame: Baseline, Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS
Population: Participants in the FAS for whom serum ferritin data were available at both Baseline and the indicated post-treatment time point. The FAS included all participants who received at least 1 complete infusion of sebelipase alfa in this study and who had at least 1 post-treatment measurement in this study.
Measure: Mean (Standard Deviation); unit: microgram (µg)/L
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
microgram (µg)/L
  Week 12 | -37.0 (29.93)
  Week 24 | -40.1 (47.27)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -18.1 (32.68)
  Week 104 | -22.8 (44.57)
  Week 156 | 0.0 (34.50)
  Week 208: number analyzed (Participants) | 7
  Week 208 | 18.0 (40.41)
  Week 260: number analyzed (Participants) | 5
  Week 260 | 63.0 (70.53)
  EOS: number analyzed (Participants) | 7
  EOS | 47.7 (56.06)

8. Secondary Outcome: Changes From Baseline In Hs-CRP
Description: Changes from Baseline to Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS for high sensitivity C-reactive protein (hs-CRP). Baseline values were defined as the last measurement prior to the first infusion of sebelipase alfa in Study LAL-CL04.
Time Frame: Baseline, Week 12, Week 24, Week 52, Week 104, Week 156, Week 208, Week 260, and EOS
Population: Participants in the FAS for whom hs-CRP data were available at both Baseline and the indicated post-treatment time point. The FAS included all participants who received at least 1 complete infusion of sebelipase alfa in this study and who had at least 1 post-treatment measurement in this study.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Open-Label Sebelipase Alfa
Number analyzed (Participants) | 8
mg/L
  Week 12 | -1.41 (3.022)
  Week 24 | -1.03 (3.945)
  Week 52: number analyzed (Participants) | 7
  Week 52 | -1.40 (3.245)
  Week 104 | -1.50 (4.079)
  Week 156 | -1.09 (3.323)
  Week 208: number analyzed (Participants) | 7
  Week 208 | -1.34 (3.674)
  Week 260: number analyzed (Participants) | 5
  Week 260 | -0.16 (0.619)
  EOS: number analyzed (Participants) | 7
  EOS | -1.33 (2.985)

ADVERSE EVENTS:
Time Frame: From after first dose administration post-Baseline through EOS during study LAL-CL04
Description: Adverse events were obtained through participant reporting or were elicited by specific questioning or examination of the participant.
Groups:
- Open-Label Sebelipase Alfa: Participants were administered sebelipase alfa qw as an IV infusion at the same dose received in Study LAL-CL01 (0.35, 1, or 3 mg/kg) for 4 weeks. After the initial 4 qw doses, participants transitioned to qow dosing at either 1 mg/kg (participants who initiated treatment at 0.35 or 1 mg/kg qw) or 3 mg/kg (participants who initiated dosing at 3 mg/kg qw). Subsequent modifications to the dose and dosing frequency were permitted for individual participants based on observed safety, tolerability, and clinical response to treatment. Participants could continue to receive treatment with sebelipase alfa for up to 5 years.
Arm/Group | Open-Label Sebelipase Alfa
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Sebelipase Alfa (N=8)
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1 — Cholecystectomy for cholelithiasis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Open-Label Sebelipase Alfa (N=8)
Bradycardia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 3
Blepharitis (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Occular hyperaemia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Faeces soft (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Malocclusion (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Catheter site pain (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Granulomatous liver disease (Hepatobiliary disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Abscess limb (Infections and infestations) | 1
Bacterial vaginosis (Infections and infestations) | 1/2 — Affects only female participants
Cellulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Ear lobe infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 5
Arthropod bite (Injury, poisoning and procedural complications) | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
Blood creatinine increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Mean cell volume increased (Investigations) | 1
Prothrombin time abnormal (Investigations) | 1
Vitamin B12 decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck mass (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Clonic convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Ephelides (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 1
Hyperaemia (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT01488097/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT01488097/SAP_001.pdf